CLINICAL TRIAL: NCT02858895
Title: An Open-Label Non-Randomized, Multi-Center Phase-2 Study of Convection-Enhanced Delivery (CED) of MDNA55 in Adults With Recurrent or Progressive Glioblastoma
Brief Title: Convection-Enhanced Delivery (CED) of MDNA55 in Adults With Recurrent or Progressive Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicenna Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDNA55-05
Record Dates: First submitted 2016-07-28; First posted 2016-08-08 (Estimated); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Glioblastoma; Grade IV Astrocytoma; Glioblastoma Multiforme; Grade IV Glioma
Keywords: High grade glioma; malignant glioma; recurrent glioblastoma; recurrent GBM; recurrent GB; glioblastoma (GB); glioblastoma multiforme (GBM); progressive glioblastoma; Brain tumor; Brain cancer; immunotherapy; targeted; IL4R
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — interleukin-4-Pseudomonas exotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDNA55 (Experimental): Single infusion of MDNA55 via convection enhanced delivery (CED).*
  *Subjects may be eligible to receive a second administration of MDNA55.
  Interventions: Drug: MDNA55

INTERVENTIONS:
Drug: MDNA55 — MDNA55 is an engineered circularly permuted interleukin-4 (cpIL-4) genetically fused to the catalytic domain of the pseudomonas exotoxin A (PE).
  Other Names: IL4-PE; Interleukin-4 Pseudomonas Exotoxin; Interleukin-4 Pseudomonas Toxin; IL4 Pseudomonas Exotoxin; NBI-3001; cpIL4-PE

SUMMARY:
This is a single-arm, open-label, multicenter study in approximately 52 adults with primary (de novo) GB that has recurred or progressed (first or second recurrence, including this recurrence) after treatment(s) including surgery and radiotherapy with or without chemotherapy and following discontinuation of any previous standard or investigational lines of therapy.

DETAILED DESCRIPTION:
The study drug, MDNA55, is a fusion protein comprising a genetically engineered Interleukin-4 (IL-4) linked to a modified version of the Pseudomonas aeruginosa exotoxin A (PE). MDNA55 binds to the IL-4 receptor (IL4R), over-expressed by cancer cells and non-malignant immunosuppressive cells of the tumor microenvironment (TME), and delivers a potent cell-killing agent, PE.

The study will be conducted at up to 10 clinical sites following institutional review board approval and completed informed consent.

Subjects that meet the study eligibility criteria will undergo surgery associated with study drug administration. MDNA55 will be administered locally by convection-enhanced delivery (CED).

Post-treatment follow-up assessment of safety and efficacy will be performed monthly for the first 6 months and bimonthly thereafter for approximately 1 year after study drug administrations. Subjects will continued to be followed for survival and post-study treatment(s) of GB after study completion or withdrawal.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subjects must be ≥ 18 years old and have a life expectancy ≥ 12 weeks
2. Histologically proven, primary (de novo) GB that has recurred or progressed (first or second recurrence, including this recurrence)
3. Confirmation that archived tissue is available from first diagnosis of GB for biomarker analysis
4. Recurrent tumor must be supratentorial, contrast-enhancing GB no smaller than 1 cm x 1 cm (largest perpendicular dimensions) and no larger than 4 cm maximum in a single direction based on MRI taken within 14 days prior to catheter placement
5. Karnofsky Performance Score (KPS) ≥ 70
6. Subjects must be able and willing to undergo multiple brain MRI examinations
7. Subjects must be able and willing to comply with all study procedures
8. Any related toxicities following discontinuation of prior GB therapies must have resolved to CTCAE Grade 1 or lower prior to inclusion in this study

EXCLUSION CRITERIA:

1. Prior treatment with cytotoxic chemotherapy

   1. Temozolomide (standard induction and / or maintenance dosing) within the past 4 weeks prior to planned infusion
   2. "Metronomic" Temozolomide (low-dose, continuous administration) within the past 7 days prior to planned infusion
   3. Nitrosoureas within the past 6 weeks prior to planned infusion
   4. Treatment with any other cytotoxic agent within the past 4 weeks prior to planned infusion
2. Prior investigational treatment within the past 4 weeks or prior immunotherapy or antibody therapy within the past 4 weeks prior to planned infusion
3. Prior treatment with bevacizumab (Avastin) or other vascular-endothelial growth factor (VEGF) inhibitors or VEGF-receptor signaling inhibitors within the past 4 weeks prior to planned infusion
4. Prior therapy that included interstitial brachytherapy or Gliadel® Wafers (carmustine implants) within the past 12 weeks prior to planned infusion
5. Prior surgery (including stereotactic radiosurgery and biopsy procedures) within the past 4 weeks prior to planned infusion
6. Ongoing Optune© therapy within 5 days of planned infusion
7. Secondary GB (i.e., GB that progressed from low-grade diffuse astrocytoma or AA)
8. Known mutation in either the isocitrate dehydrogenase 1 (IDH1) or the IDH2 gene.
9. Tumor in the brainstem (not including fluid-attenuated inversion recovery [FLAIR] changes), an infratentorial tumor, diagnosis of gliomatosis cerebri (highly infiltrative T2 hyperintense tumor with ill-defined margins encompassing at least three lobes of the brain.
10. Tumor with a mass effect (e.g. 1-2 cm midline shift)
11. Subjects with tumors for which the preponderance of tissue is not of the type in which convection would be possible (e.g. preponderance of cystic component)
12. Tumor with geometric features that make them difficult to adequately cover the tumor volume with infusate by using CED catheters
13. Clinical symptoms that are thought by the Investigator to be caused by uncontrolled increased intracranial pressure, hemorrhage, or edema of the brain
14. Any condition that precludes the administration of anesthesia
15. Known to be human immunodeficiency virus positive
16. Concurrent or a history of any significant medical illnesses that in the Investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the subject's ability to tolerate the study drug therapy and/or put the subject at additional risk or interfere with the interpretation of the results of this trial
17. Known history of allergy to gadolinium contrast agents
18. Presence of another type of malignancy requiring treatment within < 3 years prior to the screening visit, except for adequately treated carcinoma in-situ of the cervix, prostate cancer not actively treated, and basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Therapy and Research Center at The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sampson JH, Singh Achrol A, Aghi MK, Bankiewicz K, Bexon M, Brem S, Brenner A, Chandhasin C, Chowdhary S, Coello M, Ellingson BM, Floyd JR, Han S, Kesari S, Mardor Y, Merchant F, Merchant N, Randazzo D, Vogelbaum M, Vrionis F, Wembacher-Schroeder E, Zabek M, Butowski N. Targeting the IL4 receptor with MDNA55 in patients with recurrent glioblastoma: Results of a phase IIb trial. Neuro Oncol. 2023 Jun 2;25(6):1085-1097. doi: 10.1093/neuonc/noac285. PMID 36640127
- [Derived] Ellingson BM, Sampson J, Achrol AS, Aghi MK, Bankiewicz K, Wang C, Bexon M, Brem S, Brenner A, Chowdhary S, Floyd JR, Han S, Kesari S, Randazzo D, Vogelbaum MA, Vrionis F, Zabek M, Butowski N, Coello M, Merchant N, Merchant F. Modified RANO, Immunotherapy RANO, and Standard RANO Response to Convection-Enhanced Delivery of IL4R-Targeted Immunotoxin MDNA55 in Recurrent Glioblastoma. Clin Cancer Res. 2021 Jul 15;27(14):3916-3925. doi: 10.1158/1078-0432.CCR-21-0446. Epub 2021 Apr 16. PMID 33863808
- See also: Sponsor website — http://www.medicenna.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-treatment catheter trajectory planning performed to place up to 4 catheters, depending upon the tumor size.
Groups:
- MDNA55: Subjects received a single infusion of MDNA55 (via convection enhanced delivery) at concentrations ranging from 1.5 to 9.0 μg/mL. Total dose administered did not exceed 240 μg (the established maximum tolerated dose [MTD]).
Period: Overall Study
Arm/Group | MDNA55
Started | 47
Intent to Treat/Safety Population | 47 (Intent-to-Treat and Safety populations were identical and consisted of all subjects who signed an informed consent form and received any amount of study drug.)
Per Protocol Population | 44 (Per-Protocol Population consisted of all subjects in the Intent to Treat Population who had no major protocol violation during the study. Efficacy analyses were conducted on this population in support of the primary efficacy results.)
Completed | 8 (Patients who completed the study were those who completed active study follow up to Day 360)
Not Completed | 39
Not completed — Disease progression | 31
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — hospice, | 1
Not completed — did not receive drug due to catheters misplaced | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat and Safety: ITT and Safety populations were identical and consisted of all subjects who signed an informed consent form and received any amount of study drug.
Groups:
- MDNA55: Subjects received a single infusion of MDNA55 (via convection enhanced delivery) at concentrations ranging from 1.5 to 9.0 μg/mL and volumes ranging from 12 to 66 mL (total dose between 18 to 240 mcg)
Arm/Group | MDNA55
Number analyzed (Participants) | 47
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 56.7 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 2
  Native Hawaiian or Other Pacific Islander | 0
  White | 41
  Other | 3
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 44
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants]
  70 (caring for self, not capable of normal activity or work) | 3
  80 (normal activity with some difficulty, some symptoms or signs) | 20
  90 (capable of normal activity, few symptoms or signs of disease) | 19
  100 (normal, no complaints, no signs of disease) | 5
o6-methylguanine-DNA-methyltransferase (MGMT) Status [Count of Participants; unit: Participants]
  Methylated | 18
  Unmethylated | 24
  Not Available | 5
Steroid Use [Count of Participants; unit: Participants]
  Yes | 19
  No | 13
  Not applicable | 14
  Missing | 1
Diagnostic method of Glioblastoma [Number; unit: participants]
  CT | 4
  MRI | 32
  Biopsy | 30
Prior Glioblastoma treatment [Number; unit: participants]
  Initial Surgery - Total Resection | 37
  Initial Surgery - Partial Resection | 4
  Initial Surgery - Other | 6
  Additional Surgery - Resection | 10
  Additional Surgery - Debulking | 6
  Additional Surgery - Other | 4
  Radiotherapy | 46
  Temozolomide | 46
  Other Chemotherapy | 5
  Investigational | 13
  Other | 7
Initial diagnosis to 1st relapse [Mean (Standard Deviation); unit: months] | 12.98 (7.673)
Max tumor diameter at initial diagnosis [Mean (Standard Deviation); unit: cm] | 3.331 (1.4310)
Number of prior relapse [Count of Participants; unit: Participants]
  1st relapse | 37
  2nd relapse | 10
Tumor volume at baseline [Mean (Standard Deviation); unit: cm^3] | 10.543 (11.0621)
Maximum tumor diameter at baseline [Mean (Standard Deviation); unit: cm] | 3.160 (1.1736)
Lymphocyte Count [Mean (Standard Deviation); unit: 10^9 cells/L] | 0.991 (0.3839)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Primary endpoint analysis was based on the ITT population. The null hypothesis was mOS of 8.0 months, based on a clinically-weighted average of published studies of FDA-approved therapies versus the alternative hypothesis of 11.5 months.
Time Frame: From start of treatment until date of death from any cause. Subjects who were not known to have died at the time of the analysis were to be censored at the date of last contact.
Population: Primary endpoint analysis was based on the ITT population. The null hypothesis was mOS of 8.0 months, based on a clinically-weighted average of published studies of FDA-approved therapies.
  ITT/Safety population: all subjects who signed an informed consent form and received any amount of study drug.
  Per-Protocol Population: all subjects in the ITT Population who had no major protocol violation during the study.
  Primary efficacy analysis was not performed for individual dose concentrations.
Measure: Median (80% Confidence Interval); unit: months
Groups:
- MDNA55 (ITT Analysis): All subjects enrolled, received any amount of study drug
- MDNA55 (PP Analysis): In support of the primary efficacy analysis, evaluation of the primary endpoint was also conducted on the PP population.
Arm/Group | MDNA55 (ITT Analysis) | MDNA55 (PP Analysis)
Number analyzed (Participants) | 47 | 44
months | 10.2 [8.39 to 12.75] | 11.64 [8.62 to 15.02]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR, determined by independent central review (per RANO-based criteria) Complete Response - Disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks.
  Partial Response - ≥50% decrease in sum of products of perpendicular diameters or ≥65% decrease in total volume of all measurable enhancing lesions compared with baseline, sustained for at least 4 weeks Progressive Disease - At least two sequential scans separated by at ≥4 weeks both exhibiting ≥25% increase in sum of products of perpendicular diameters or ≥40% increase in total volume of enhancing lesions.
  Stable Disease - Does not qualify for CR, PR, or PD as defined above
Time Frame: 12 months
Population: Modified Intent-to-Treat Population (mITT): mITT population was used for secondary response analyses and consisted of all subjects who received any amount of study drug, had adequate imaging (at least 1 post-treatment scan), and had sufficient clinical data for ORR analysis.
Measure: Count of Participants; unit: Participants
Groups:
- MDNA55: Single infusion of MDNA55 via convection enhanced delivery (CED).*
  *Subjects may be eligible to receive a second administration of MDNA55.
  MDNA55: MDNA55 is an engineered circularly permuted interleukin-4 (cpIL-4) genetically fused to the catalytic domain of the pseudomonas exotoxin A (PE).
Arm/Group | MDNA55
Number analyzed (Participants) | 41
Participants | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, time from treatment until disease progression (per RANO-based criteria) or death Progressive Disease per RANO - At least two sequential scans separated by at ≥4 weeks both exhibiting ≥25% increase in sum of products of perpendicular diameters or ≥40% increase in total volume of enhancing lesions
Time Frame: 12 months
Population: as for outcome 2
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | MDNA55
Number analyzed (Participants) | 41
months | 3.61 [2.79 to 5.08]

4. Other Pre Specified Outcome: Number of Subjects With Serious Adverse Events
Description: Number of Subjects with Serious adverse events with Frequency >=5%
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- MDNA55: Single infusion of MDNA55 via convection enhanced delivery (CED).
  MDNA55: MDNA55 is an engineered circularly permuted interleukin-4 (cpIL-4) genetically fused to the catalytic domain of the pseudomonas exotoxin A (PE).
Arm/Group | MDNA55
Number analyzed (Participants) | 47
Participants | 24

5. Other Pre Specified Outcome: Treatment Emergent Adverse Events
Description: Incidence of Treatment-Emergent adverse events
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MDNA55
Number analyzed (Participants) | 47
Participants | 46

6. Other Pre Specified Outcome: Level of MDNA55 in Peripheral Plasma
Description: Systemic exposure to MDNA55 is not expected following intratumoral infusion and circulating MDNA55 has not been detected in previous clinical studies. To continue to evaluate the potential of systemic exposure, plasma collected at screening (baseline), within 1 hour following infusion end time, ~3 hours following completion of infusion and then (after the ~3 hour sample collection) every 6 hours ± 2 hours until 24 hours and at Day 14. PK data will be presented for the PK population in listing format by subject and sample collection time point. PK parameters would only be analyzed if MDNA55 levels above LLOQ (0.37 ng/mL) were detected.
Time Frame: 14 days
Population: Pharmacokinetic (PK) Population: Subjects who received the highest concentrations (6 μg/mL and 9 μg/mL) were analysed first. If all results were shown to be below lower limit of quantitation (LLOQ) of 0.37 ng/mL, consistent with historical data showing no evidence of systemic exposure with MDNA55, then no further subjects were to be analyzed. All subjects analyzed had levels of MDNA55 that were below lower limit of quantitation (LLOQ) of 0.37 ng/mL
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | MDNA55
Number analyzed (Participants) | 28
ng/mL | NA (NA) — All MDNA55 levels below LLOQ

7. Other Pre Specified Outcome: ADA Titer / Neutralizing Antibody Analysis
Description: Number of participants that were ADA Positive and had Neutralizing Antibody
Time Frame: 12 months
Population: Anti-Drug-Antibody (ADA) Population: ADA population included all subjects who received any dose of study drug and had a pre-treatment baseline blood sample and at least one post-treatment blood sample available for determination of ADA. Neutralizing antibody (NAb) titers were assessed in the ADA population as appropriate and applicable.
Measure: Count of Participants; unit: Participants
Arm/Group | MDNA55
Number analyzed (Participants) | 46
Participants
  ADA positive | 19
  Neutralizing Antibody (NAb): number analyzed (Participants) | 19
  Neutralizing Antibody (NAb) | 16

ADVERSE EVENTS:
Time Frame: AEs were collected from catheter placement through 12 months post treatment or early withdrawal and followed until resolution, stabilization, data cut-off, or death. For subjects that withdraw from the study, SAEs that occur within 30 days of the date of discontinuation collected.
Description: All patients were included in the in the ITT / Safety Population (N=47) for "MDNA55 (Overall)"; there is one patient that underwent catheter placement but did not receive the study drug; the infusion did not proceed due to catheter misplacement. Therefore, this participant is not included in the individual MDNA55 infusion arms (N=46)
Groups:
- MDNA55 (Overall): Single infusion of MDNA55 administered via Convection Enhanced Delivery (CED) Dose conc. range 1.5 to 9.0 mcg/mL; total dose range 18 to 240 mcg
- MDNA55 (1.5 mcg/mL): Single infusion of MDNA55 administered via Convection Enhanced Delivery (CED) Dose conc. 1.5 mcg/mL
- MDNA55 (3.0 mcg/mL): Single infusion of MDNA55 administered via Convection Enhanced Delivery (CED) Dose conc. 3.0 mcg/mL
- MDNA55 (6.0 mcg/mL): Single infusion of MDNA55 administered via Convection Enhanced Delivery (CED) Dose conc. 6.0 mcg/mL
- MDNA55 (9.0 mcg/mL): Single infusion of MDNA55 administered via Convection Enhanced Delivery (CED) Dose conc. 9.0 mcg/mL
Arm/Group | MDNA55 (Overall) | MDNA55 (1.5 mcg/mL) | MDNA55 (3.0 mcg/mL) | MDNA55 (6.0 mcg/mL) | MDNA55 (9.0 mcg/mL)
All-Cause Mortality (participants affected / at risk) | 36/47 | 16/18 | 8/9 | 3/6 | 8/13
Serious Adverse Events (participants affected / at risk) | 24/47 | 7/18 | 4/9 | 3/6 | 9/13
Other Adverse Events (participants affected / at risk) | 46/47 | 18/18 | 9/9 | 6/6 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDNA55 (Overall) (N=47) | MDNA55 (1.5 mcg/mL) (N=18) | MDNA55 (3.0 mcg/mL) (N=9) | MDNA55 (6.0 mcg/mL) (N=6) | MDNA55 (9.0 mcg/mL) (N=13)
Seizure (Nervous system disorders) | 8 (9) | 4 (5) | 1 (1) | 2 (2) | 1 (1)
Brain oedema (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication of Device Insertion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neurological Decompensation (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neurological Symptom (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritumoral Oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDNA55 (Overall) (N=47) | MDNA55 (1.5 mcg/mL) (N=18) | MDNA55 (3.0 mcg/mL) (N=9) | MDNA55 (6.0 mcg/mL) (N=6) | MDNA55 (9.0 mcg/mL) (N=13)
Agitation (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (6) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 12 (18) | 4 (4) | 3 (4) | 2 (5) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Blood albumin decreased (Investigations) | 2 (5) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (5) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 2 (4) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Brain oedema (Nervous system disorders) | 5 (6) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
Cognitive disorder (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 7 (7) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 4 (6) | 2 (3) | 1 (1) | 1 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Extensor plantar response (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Facial paresis (Nervous system disorders) | 7 (7) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 19 (23) | 8 (9) | 3 (5) | 3 (4) | 5 (5)
Gait disturbance (General disorders) | 7 (10) | 0 (0) | 3 (3) | 1 (4) | 3 (3)
Headache (Nervous system disorders) | 18 (35) | 10 (10) | 2 (7) | 4 (13) | 2 (5)
Hemiparesis (Nervous system disorders) | 12 (17) | 4 (4) | 2 (2) | 1 (4) | 5 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (5) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (13) | 1 (1) | 4 (4) | 4 (5) | 3 (3)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (13) | 3 (10) | 1 (2) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 5 (6) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 (18) | 8 (9) | 1 (1) | 1 (2) | 5 (6)
Nausea (Gastrointestinal disorders) | 8 (10) | 3 (3) | 2 (3) | 1 (2) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 7 (7) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Partial seizures (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 8 (17) | 1 (2) | 1 (1) | 3 (9) | 3 (5)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 14 (17) | 4 (5) | 2 (2) | 5 (7) | 3 (3)
Simple partial seizures (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Vision blurred (Eye disorders) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (8) | 2 (2) | 2 (3) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02858895/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT02858895/SAP_001.pdf